CLINICAL TRIAL: NCT05066360
Title: Investigation of Serum Antimullerian Hormone Levels in Adolescent Epilepsy Patients
Brief Title: Serum Antimullerian Hormone Levels Among Epileptic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Ali Cenk, Medical Doctor, Associate Professor, Near East University, Turkey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AMH
Record Dates: First submitted 2021-07-02; First posted 2021-10-04 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Epilepsy; Reproductive Issues
Keywords: anti-mullerian hormone; epilepsy; adolescent
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: two groups (epileptic and healthy participants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- participants with epilepsy (Other): healthy, menstruating females between 12-18 ages
  Interventions: Diagnostic Test: serum antimullerian hormone
- healthy participants (Other): epileptic, menstruating females between 12-18 ages
  Interventions: Diagnostic Test: serum antimullerian hormone

INTERVENTIONS:
Diagnostic Test: serum antimullerian hormone — serum antimullerian hormone will be analyzed for all participants

SUMMARY:
The production of AMH starts in granulosa cells before birth and the levels within the serum decreases towards the menapouse. The levels of AMH do not change throughout the menstruation cycle hovewer, it can be affected in cases related to body mass index (BMI), polycyctic ovarian syndrome (PCOS). The lower levels of AMH had been documented after ovarian surgery, radiotheraphy and chemotheraphy. AMH is a member of Transforming Growth Faktor β (TGF- β ) and it has receptors in brain structures including hyppocammpus. It is highly active neurophysiologically and it has a protective effect against N-methyl-D -aspartate related neuronal injury that is demonstrated both in vivo and in vitro studies. As a result, being a neuroactive hormone; AMH may have an effect on seizures within epileptic patients or serum AMH levels may be effected in epileptic patients when compared with healthy ones.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and epileptic volunteer females
* Ages between 12-18
* After menarche

Exclusion Criteria:

* ovarian surgery,
* history of radiotherapy
* history of chemotherapy,
* before menarche

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
serum anti-mullerian hormone levels | baseline, at the time of examination
  The comparison of serum levels of anti-mullerian hormone between epileptic and healthy groups

CONTACTS AND LOCATIONS:
Overall Officials: ALİ ÖZAY, Assoc Prof, Principal Investigator — Near East University
Locations (1):
- Near East University Faculty of Medicine, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No
Serum antimullerian hormone levels will be shared for both groups

REFERENCES:
- [Background] Karkanaki A, Vosnakis C, Panidis D. The clinical significance of anti-Mullerian hormone evaluation in gynecological endocrinology. Hormones (Athens). 2011 Apr-Jun;10(2):95-103. doi: 10.14310/horm.2002.1299. PMID 21724534
- [Background] Practice Committee of the American Society for Reproductive Medicine. Testing and interpreting measures of ovarian reserve: a committee opinion. Fertil Steril. 2015 Mar;103(3):e9-e17. doi: 10.1016/j.fertnstert.2014.12.093. Epub 2015 Jan 10. PMID 25585505
- [Background] Visser JA, de Jong FH, Laven JS, Themmen AP. Anti-Mullerian hormone: a new marker for ovarian function. Reproduction. 2006 Jan;131(1):1-9. doi: 10.1530/rep.1.00529. PMID 16388003
- [Background] Cimino I, Casoni F, Liu X, Messina A, Parkash J, Jamin SP, Catteau-Jonard S, Collier F, Baroncini M, Dewailly D, Pigny P, Prescott M, Campbell R, Herbison AE, Prevot V, Giacobini P. Novel role for anti-Mullerian hormone in the regulation of GnRH neuron excitability and hormone secretion. Nat Commun. 2016 Jan 12;7:10055. doi: 10.1038/ncomms10055. PMID 26753790
- [Background] Lebeurrier N, Launay S, Macrez R, Maubert E, Legros H, Leclerc A, Jamin SP, Picard JY, Marret S, Laudenbach V, Berger P, Sonderegger P, Ali C, di Clemente N, Vivien D. Anti-Mullerian-hormone-dependent regulation of the brain serine-protease inhibitor neuroserpin. J Cell Sci. 2008 Oct 15;121(Pt 20):3357-65. doi: 10.1242/jcs.031872. Epub 2008 Sep 16. PMID 18796535
- [Background] Harden CL, Pennell PB. Neuroendocrine considerations in the treatment of men and women with epilepsy. Lancet Neurol. 2013 Jan;12(1):72-83. doi: 10.1016/S1474-4422(12)70239-9. PMID 23237902
- [Background] Harden CL, Koppel BS, Herzog AG, Nikolov BG, Hauser WA. Seizure frequency is associated with age at menopause in women with epilepsy. Neurology. 2003 Aug 26;61(4):451-5. doi: 10.1212/01.wnl.0000081228.48016.44. PMID 12939416
- [Background] Meo R, Bilo L, Nappi C, Tommaselli AP, Valentino R, Nocerino C, Striano S, Buscaino GA. Derangement of the hypothalamic GnRH pulse generator in women with epilepsy. Seizure. 1993 Sep;2(3):241-52. doi: 10.1016/s1059-1311(05)80134-7. PMID 8162389
- [Background] Herzog AG, Coleman AE, Jacobs AR, Klein P, Friedman MN, Drislane FW, Ransil BJ, Schomer DL. Interictal EEG discharges, reproductive hormones, and menstrual disorders in epilepsy. Ann Neurol. 2003 Nov;54(5):625-37. doi: 10.1002/ana.10732. PMID 14595652
- [Background] Quigg M, Kiely JM, Johnson ML, Straume M, Bertram EH, Evans WS. Interictal and postictal circadian and ultradian luteinizing hormone secretion in men with temporal lobe epilepsy. Epilepsia. 2006 Sep;47(9):1452-9. doi: 10.1111/j.1528-1167.2006.00617.x. PMID 16981860
- [Background] Harden CL, Pennell PB, French JA, Davis A, Lau C, Llewellyn N, Kaufman B, Bagiella E, Kirshenbaum A. Anti-mullerian hormone is higher in seizure-free women with epilepsy compared to those with ongoing seizures. Epilepsy Res. 2016 Nov;127:66-71. doi: 10.1016/j.eplepsyres.2016.08.003. Epub 2016 Aug 17. PMID 27565413